CLINICAL TRIAL: NCT02132806
Title: Piezosurgery in the Treatment of Class II Furcation Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Matteo Visintin (Other)
Responsible Party: Sponsor-Investigator, Matteo Visintin, Student, University of Trieste
Organization: University of Trieste (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNITS01-2014
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Furcation Defects
Keywords: class II furcation involvement; piezoelectric surgery; regeneration; biomaterial
MeSH Terms: conditions — Furcation Defects | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OFD with piezosurgery (Experimental): Open flap debridement with Piezosurgery
  Interventions: Procedure: Piezosurgery
- OFD with piezosurgery+biomaterial (Experimental): Open flap debridement with Piezosurgery with biomaterial mp3
  Interventions: Procedure: Piezosurgery with biomaterial mp3
- OFD with piezosurgery+mp3+bracket (Experimental): Open flap debridement with Piezosurgery with biomaterial mp3 + bracket
  Interventions: Procedure: Piezosurgery with biomaterial mp3 + bracket

INTERVENTIONS:
Procedure: Piezosurgery with biomaterial mp3 + bracket
  Arms: OFD with piezosurgery+mp3+bracket
Procedure: Piezosurgery with biomaterial mp3
  Arms: OFD with piezosurgery+biomaterial
Procedure: Piezosurgery
  Arms: OFD with piezosurgery

SUMMARY:
The purpose of this study is to evaluate the effectiveness of piezosurgery in the treatment of class II furcation involvement using biomaterials and new surgical techniques

ELIGIBILITY:
Inclusion Criteria:

* previous subgingival instrumentation with adequate plaque control (FMPS < 20%) and bleeding on probing (FMBS < 20%).
* one or more mandibular molar with buccal class-II furcation involvement

Exclusion Criteria:

* diabetes mellitus
* pregnancy and lactation period
* subjects smoking > 10 cigarettes/day were excluded
* subjects in chronically treatment with calcium antagonist, immunosuppressive drugs and Antiepileptic Drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Horizontal probing depth (PH) | 180 days
  horizontal probing depth

SECONDARY OUTCOMES:
Plaque index (PI) | 180 days
  plaque index
Bleeding on probing (BoP) | 180 days
  bleeding on probing
Pocket probing depth (PPD) | 180 days
  pocket probing depth
Furcation closure (FC) | 180 days
  furcation closure
Clinical attachment level (CAL) | 180 days
  clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Visintin, Principal Investigator — UCO Clinica Odontoiatrica e Stomatologica - Ospedale Maggiore Trieste
Locations (1):
- Matteo Visintin, Trieste, TS, Italy